CLINICAL TRIAL: NCT00405522
Title: Co-administration of Propofol and Remifentanil for Lumbar Puncture in Children: Evaluation of Two Dose Combinations
Brief Title: Co-administration of Propofol and Remifentanil for Lumbar Puncture in Children
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Jason Hayes, Staff Anesthesiologist, The Hospital for Sick Children
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1000009427
Record Dates: First submitted 2006-11-28; First posted 2006-11-30 (Estimated); Results first posted 2019-03-08 (Actual); Last update posted 2019-03-08 (Actual); Status verified 2018-11

CONDITIONS: Spinal Puncture
Keywords: Lumbar Puncture; Pediatrics; Propofol; Remifentanil; sedation; Oncology
MeSH Terms: conditions — Neoplasms | interventions — Propofol; Remifentanil

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Propofol 2.0 mg/kg + Remifentanil 1.5 ug/kg (Experimental)
  Interventions: Drug: Propofol 2.0 mg/kg + Remifentanil 1.5 ug/kg
- Propofol 4.0 mg/kg + Remifentanil 0.5 ug/kg (Experimental)
  Interventions: Drug: Propofol 4.0 mg/kg + Remifentanil 0.5 ug/kg

INTERVENTIONS:
Drug: Propofol 2.0 mg/kg + Remifentanil 1.5 ug/kg — Patients in this arm of the study will receive 2.0 mg/kg propofol + 1.5 ug/kg remifentanil. An anesthesiologist will inject propofol mixed with lidocaine, followed immediately by remifentanil, diluted with 0.9% saline to a volume of 3 ml and administered as a bolus.
  Arms: Propofol 2.0 mg/kg + Remifentanil 1.5 ug/kg
Drug: Propofol 4.0 mg/kg + Remifentanil 0.5 ug/kg — Patients in this arm of the study will receive 4.0 mg/kg propofol + 0.5 ug/kg remifentanil. An anesthesiologist will inject propofol mixed with lidocaine, followed immediately by remifentanil, diluted with 0.9% saline to a volume of 3 ml and administered as a bolus.
  Arms: Propofol 4.0 mg/kg + Remifentanil 0.5 ug/kg

SUMMARY:
The objective of this study is to compare intraoperative and recovery parameters in patients who receive two different dose combinations of propofol and remifentanil in patients undergoing a lumbar puncture.

DETAILED DESCRIPTION:
Lumbar punctures (LP) are performed in approximately one thousand oncology patients per year at the Hospital for Sick Children. In a previous study, we determined the optimal dose of remifentanil which provides effective anesthesia with little or no movement during LP in children. The present study will determine the optimal dose combination of propofol and remifentanil to keep patients comfortable and still during the procedure while decreasing the incidence of side effects and allows for shorter recovery times and earlier discharge from the recovery room.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of a hemato-oncological disorder
* Scheduled to undergo a lumbar puncture
* Aged 3-12 years
* Unpremedicated

Exclusion Criteria:

* children who are known or suspected to be difficult to ventilate by face mask
* children who are deemed medically unfit to receive either of the two study medications
* children who are obese (weight for height > 95th percentile)
* children who do not have an indwelling intravenous line

Ages: 3 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 34 (Actual)
Dates: Start 2006-11; Primary Completion 2007-06 (Actual); Study Completion 2007-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jason Hayes, MD, Principal Investigator — The Hospital for Sick Children, Toronto Canada
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada

RESULTS

PARTICIPANT FLOW:
Groups:
- 2.0 mg/kg Propofol: Propofol + Remifentanil: Patients in this arm of the study will receive 2.0 mg/kg propofol + 1.5 ug/kg remifentanil. An anesthesiologist will inject propofol mixed with lidocaine, followed immediately by remifentanil, diluted with 0.9% saline to a volume of 3 ml and administered as a bolus.
- 4.0 mg/kg Propofol: Propofol + Remifentanil: Patients in this arm of the study will receive 4.0 mg/kg propofol + 0.5 ug/kg remifentanil. An anesthesiologist will inject propofol mixed with lidocaine, followed immediately by remifentanil, diluted with 0.9% saline to a volume of 3 ml and administered as a bolus.
Period: Overall Study
Arm/Group | 2.0 mg/kg Propofol | 4.0 mg/kg Propofol
Started | 17 | 17
Completed | 17 | 17
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- 2.0 mg/kg Propofol and 1.5 ug/kg Remifentanil: Propofol + Remifentanil: Patients in this arm of the study will receive 2.0 mg/kg propofol + 1.5 ug/kg remifentanil. An anesthesiologist will inject propofol mixed with lidocaine, followed immediately by remifentanil, diluted with 0.9% saline to a volume of 3 ml and administered as a bolus.
- 4.0 mg/kg Propofol and 0.5 ug/kg Remifentanil: Propofol + Remifentanil: Patients in this arm of the study will receive 4.0 mg/kg propofol + 0.5 ug/kg remifentanil. An anesthesiologist will inject propofol mixed with lidocaine, followed immediately by remifentanil, diluted with 0.9% saline to a volume of 3 ml and administered as a bolus.
- Total: Total of all reporting groups
Arm/Group | 2.0 mg/kg Propofol and 1.5 ug/kg Remifentanil | 4.0 mg/kg Propofol and 0.5 ug/kg Remifentanil | Total
Number analyzed (Participants) | 17 | 17 | 34
Age, Continuous [Mean (Standard Deviation); unit: years] | 6.2 (1.6) | 7.2 (2.4) | 6.6 (2.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 15 | 19
  Male | 13 | 2 | 15

OUTCOME MEASURES:

1. Primary Outcome: Duration of Apnea
Description: Duration of no respiratory effort
Time Frame: This outcome was measured for the duration of the procedure (lumbar puncture).
Measure: Median (Full Range); unit: seconds
Arm/Group | 2.0 mg/kg Propofol | 4.0 mg/kg Propofol
Number analyzed (Participants) | 17 | 17
seconds | 110 [0 to 228] | 73 [0 to 110]

2. Primary Outcome: Duration of Postoperative Recovery (Time to Spontaneous Eye Opening, Verbalization, Purposeful Movement).
Time Frame: This outcome was measured for the duration of the recovery phase.
Measure: Median (Full Range); unit: minutes
Arm/Group | 2.0 mg/kg Propofol | 4.0 mg/kg Propofol
Number analyzed (Participants) | 17 | 17
minutes | 10 [4 to 70] | 23 [5 to 69]

3. Secondary Outcome: Incidence of Adverse Events and Clinically Significant Changes in Routine Vital Signs as Measured by Electrocardiogram, Non-invasive Blood Pressure, and Pulse Oximeter.
Time Frame: This outcome was measured for the duration of the procedure (lumbar puncture).
Measure: Count of Participants; unit: Participants
Arm/Group | 2.0 mg/kg Propofol | 4.0 mg/kg Propofol
Number analyzed (Participants) | 17 | 17
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were observed from the injection of study drugs until discharge from recovery room.
Groups:
- 4.0 mg/kg Propofol + 0.5 ug/kg Remifentanil: Propofol + Remifentanil: Patients in this arm of the study will receive 4.0 mg/kg propofol + 0.5 ug/kg remifentanil. An anesthesiologist will inject propofol mixed with lidocaine, followed immediately by remifentanil, diluted with 0.9% saline to a volume of 3 ml and administered as a bolus.
Arm/Group | 2.0 mg/kg Propofol and 1.5 ug/kg Remifentanil | 4.0 mg/kg Propofol + 0.5 ug/kg Remifentanil
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/17
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/17
Other Adverse Events (participants affected / at risk) | 0/17 | 0/17

LIMITATIONS AND CAVEATS:
Small sample sizes

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes